CLINICAL TRIAL: NCT02281188
Title: Registry for Treatment of Upper Urinary Tract Tumours; A Multi-Center, International Registry to Evaluate the Treatment of Upper Tract Urothelial Cancer: Incidence, Indications, Treatment Types and Outcomes.
Brief Title: Registry for Treatment of Upper Urinary Tract Tumours
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Other Study IDs: Registry UTUC
Record Dates: First submitted 2014-09-26; First posted 2014-11-03 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Upper Urinary Tract Tumours

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this registry is to evaluate the incidence, indications and outcomes of patients presenting with UTUC in relation to the different treatment modalities used.

DETAILED DESCRIPTION:
This is an observational international multi-center study in which data on consecutive patients with UUT tumours are collected. Centers from every continent may apply for participation in this registry. Data will be collected from consecutive patients over a five year period. Patients' data at baseline visit, at one year, three years and five years after inclusion in the registry will be recorded, as well as data on intra- and postoperative complications, recurrence and survival in the whole study period. Data from all participating centers will be collected through electronic case report forms (eCRFs), with use of an online Data Management System (DMS), which is located and maintained at the CROES Office.

ELIGIBILITY:
Inclusion Criteria:

* Is presenting with a suspected primary UTUC (any stage)
* Is scheduled for treatment of UUT tumour
* Has signed informed consent

Exclusion Criteria:

* No specific exclusion criteria are defined.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises those patients presenting with (a) (suspected) primary UUT tumour(s) and are planned to undergo either nephroureterectomy, ureteroscopic diagnostics and/or ureteroscopic treatment, percutaneous treatment or adjuvant treatment in the participating centers.
Sampling Method: Probability Sample
Enrollment: 2451 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence rates for patients presenting with primary UTUC stratified for type of treatment | 10 years
  Data collection will be divided into the following categories: Patient / tumour characteristics, assessment, treatment choice and intra-operative details, post-operative details and complications, and follow up. The following lists all categories and type of data to be gathered.
  Patient characteristics: demographics, risk factors, comorbidities and previous malignancies.
  Assessment: symptoms, imaging type, cytology, TNM staging. Treatment choice and intra-operative details: date, use of endoscopy, type of scopes, type of imaging enhancement, biopsies, results, neo adjuvant treatment specifications and treatment type.
  Intra-operative: date, duration, antibiotics, type of treatment, results. Post-operative: complications and Clavien-Dindo classification, instillation, adjuvant therapy, pathology.
  Follow up: date, status (e.g. alive without cancer, alive with cancer), recurrence, diagnostics performed, cystoscopy, cytology, results.

SECONDARY OUTCOMES:
Intra- and postoperative complications (including Clavien-Dindo classification) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean de la Rosette, Study Chair — Clinical Research Office of the Endourological Society
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

REFERENCES:
- [Derived] Zhao H, Liu K, Crisci A, Te Slaa E, Habuchi T, Akand M, Ng CF, Laguna P, Teoh JY, de la Rosette J. Impact of smoking status at diagnosis on oncological outcomes of upper-tract urothelial carcinoma. Ther Adv Urol. 2025 Jun 28;17:17562872251352049. doi: 10.1177/17562872251352049. eCollection 2025 Jan-Dec. PMID 40584958
- [Derived] Liu K, Leung DK, Wong CH, Ko IC, Horuz R, Gontero P, Laguna P, de la Rosette J, Teoh JY. Influence of tumour location on the survival outcomes of upper tract urothelial carcinoma treated with radical nephroureterectomy. World J Urol. 2025 May 3;43(1):261. doi: 10.1007/s00345-024-05432-0. PMID 40317391
- [Derived] Liu K, Wong CH, Zhao H, Ng CF, Teoh JY, Laguna P, de la Rosette J. Impact of Antiaggregant and Anticoagulant Medications on Perioperative Complications in Upper Tract Urothelial Carcinoma. Eur Urol Open Sci. 2025 Mar 20;75:1-6. doi: 10.1016/j.euros.2025.02.007. eCollection 2025 May. PMID 40206439
- [Derived] Baard J, Cormio L, Dasgupta R, Maruzzi D, Rais-Bahrami S, Serrano A, Geavlete B, Giannakopoulos S, de la Rosette J, Laguna P. Unveiling the challenges of UTUC biopsies and cytology: insights from a global real-world practice study. World J Urol. 2024 Mar 20;42(1):177. doi: 10.1007/s00345-024-04866-w. PMID 38507109
- [Derived] Baard J, Shariat SF, Roupret M, Yoshida T, Saita A, Saltirov I, Burgos JR, Celik O, de la Rosette J, Laguna P. Adherence to guideline recommendations in the management of upper tract urothelial carcinoma: an analysis of the CROES-UTUC registry. World J Urol. 2022 Nov;40(11):2755-2763. doi: 10.1007/s00345-022-04168-z. Epub 2022 Oct 5. PMID 36197507
- [Derived] Baard J, Cormio L, Cavadas V, Alcaraz A, Shariat SF, de la Rosette J, Laguna MP. Contemporary patterns of presentation, diagnostics and management of upper tract urothelial cancer in 101 centres: the Clinical Research Office of the Endourological Society Global upper tract urothelial carcinoma registry. Curr Opin Urol. 2021 Jul 1;31(4):354-362. doi: 10.1097/MOU.0000000000000899. PMID 34009177
- [Derived] Baard J, Celebi M, de la Rosette J, Alcaraz A, Shariat S, Cormio L, Cavadas V, Laguna MP. Evaluation of Patterns of Presentation, Practice, and Outcomes of Upper Tract Urothelial Cancer: Protocol for an Observational, International, Multicenter, Cohort Study by the Clinical Research Office of the Endourology Society. JMIR Res Protoc. 2020 Jan 24;9(1):e15363. doi: 10.2196/15363. PMID 32012106
- See also: Related Info — http://www.croesoffice.org